CLINICAL TRIAL: NCT02321891
Title: Optimizing Transcranial Electrical Stimulation for Clinical Applications (the OptES Study): A Pilot Study to Determine a Candidate Protocol for Treatment of Anxiety (OptES-Anx)
Brief Title: A Pilot Study to Determine a Candidate Protocol for Transcranial Electrical Stimulation in the Treatment of Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Soili Lehto, Adjunct professor, University of Eastern Finland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OptES-Anx-pilot
Record Dates: First submitted 2014-12-09; First posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment 1 (Experimental): NeuroConn DC Stimulator Plus, tDCS treatment protocol no 1
  Interventions: Device: NeuroConn DC Stimulator Plus, tDCS
- Treatment 2 (Experimental): NeuroConn DC Stimulator Plus, tDCS treatment protocol no 2
  Interventions: Device: NeuroConn DC Stimulator Plus, tDCS

INTERVENTIONS:
Device: NeuroConn DC Stimulator Plus, tDCS — transcranial electrical stimulation intervention with two experimental protocols

SUMMARY:
The investigators examine the efficacy of two different transcranial direct current stimulation (tDCS) stimulation protocols in the treatment of anxiety in an open-label pilot study.

DETAILED DESCRIPTION:
The investigators examine the efficacy of two different transcranial direct current stimulation (tDCS) stimulation protocols in the treatment of anxiety in an open-label pilot study in patients with chronic pain. The investigators also seek to detect autonomic nervous system changes induced by the tDCS, and develop new methods for the measurement of autonomic nervous system functions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Naïve to tDCS
* Right-handed
* Beck Anxiety Scores >= 26

Exclusion Criteria:

* Metal implants inside skull or eye
* Severe skin lesions at the electrode placement area
* History of epilepsy or previous seizures
* Pregnant or breast-feeding
* Pacemaker
* History of intracerebral bleeding during the past six months
* Lifetime DSM-IV diagnosis of bipolar mood disorder or psychotic disorder
* DSM-IV diagnosis for substance abuse or dependence during the past six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Beck Anxiety Inventory | 12 days
  change in scores of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Soili M Lehto, MD, PhD, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, Finland